CLINICAL TRIAL: NCT02513316
Title: Microbleeds and Genetic Risk Factors to Predict the Risk of Intracranial Haemorrhage in Patients Treated With Anticoagulation Following Cardioembolic Stroke Due to Atrial Fibrillation
Brief Title: Clinical Relevance of Microbleeds In Stroke
Acronym: CROMIS-2
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 11/0116
Record Dates: First submitted 2015-07-29; First posted 2015-07-31 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Stroke; Atrial Fibrillation (AF); Intracerebral Haemorrhage (ICH)
Keywords: Microbleeds
MeSH Terms: conditions — Stroke; Atrial Fibrillation; Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study I (AF): Prospective cohort study of patients anticoagulated after cardioembolic stroke started on best practice oral anticoagulant (without prior use) for presumed cardioembolic ischaemic stroke due to non-valvular AF with follow up for the occurrence of ICH, ischaemic stroke and cognitive function for an average of two years. Our main baseline exposures (risk factors of interest) are the presence of CMBs on MRI, and genetic polymorphisms in candidate genes with potential functional relevance to ICH risk.
- Study II (ICH): Observational and genetics study of intracerebral haemorrhage Patients with ICH (non anticoagulant-related ICH cases and anticoagulant-related ICH cases).

SUMMARY:
Study I: CROMIS-2 (AF) Prospective cohort study of patients anticoagulated after cardioembolic stroke An observational inception cohort study (n=1425) of patients throughout the United Kingdom (UK) - (79 hospitals) started on best practice oral anticoagulant (without prior use) for presumed cardioembolic ischaemic stroke due to non-valvular AF with follow up for the occurrence of intracerebral haemorrhage (ICH) and ischaemic stroke for an average of two years. The main baseline exposures (risk factors of interest) are the presence of cerebral microbleeds (CMBs) on magnetic resonance imaging (MRI), and genetic polymorphisms in candidate genes with potential functional relevance to ICH risk.

Study II: CROMIS-2 (ICH) Observational and genetics study of intracerebral haemorrhage The investigators will also recruit 600 patients admitted to participating centres with ICH (with a target of at least 300 anticoagulant-related ICH cases) and collect DNA to increase the power of the genetic studies. The investigators will collect clinical and imaging data from these ICH cases to investigate risk factors associated with anticoagulant-related ICH compared to non anticoagulant-related ICH.

DETAILED DESCRIPTION:
Background Over the last decade, increasing use of oral anticoagulants to prevent cardioembolic ischaemic stroke due to atrial fibrillation (AF) in an ageing population has led to a five-fold increase in the incidence of anticoagulant-related intracranial haemorrhage (ICH) - a rare but unpredictable and catastrophic complication. Cerebral microbleeds (CMBs) on magnetic resonance imaging (MRI) may predict ICH risk, as may genetic polymorphisms influencing brain small-vessel integrity or anticoagulation stability.

Aims To establish the value of CMBs and genetic factors in predicting symptomatic ICH following best practice oral anticoagulation to prevent recurrent ischaemic stroke due to AF.

Methods CROMIS-2: Study I (AF) - Prospective, multicentre, inception cohort study in 1425 patients with ischaemic stroke due to AF started on best practice oral anticoagulation. Patients will have genetic testing and standardized MRI including Gradient recalled Echo (GRE) at baseline, with follow-up by postal questionnaire (and clinical assessment or medical records surveillance after suspected events), and where possible there will be an in person clinical assessment at 2 years. The investigators will compare the rate of symptomatic ICH between CMB and CMB-free patients and test for associations with plausible candidate genes. The investigators aim to develop and validate a risk model to predict symptomatic ICH following best practice oral anticoagulation to prevent recurrent ischaemic stroke due to AF.

CROMIS-2: Study II (ICH) - An observational study of ICH investigating genetic, clinical and radiological risk factors associated with anticoagulant-related ICH. The investigators will recruit patients admitted to participating centres with ICH (with a target of at least 300 anticoagulant-related ICH cases) and collect DNA to increase the power of the genetic studies. The investigators will collect clinical and imaging data from these ICH cases to investigate risk factors associated with anticoagulant-related ICH compared to non anticoagulant-related ICH.

Expected outcomes A successful predictive model for ICH risk after best practice oral anticoagulation for AF will help to determine whether genetic or CMB screening should be used in clinical practice and future trials. New genetic, clinical and radiological risk factors associated with anticoagulant-related ICH will be identified.

ELIGIBILITY:
Study I: CROMIS-2 (AF)

Inclusion criteria:

* Adult (≥18y; no upper limit) patients with a clinical diagnosis of non-valvular AF (verified by ECG) with intention to treat with best practice oral anticoagulants (e.g. warfarin)
* Previous ischaemic stroke or TIA diagnosed by treating clinician
* All patients must be able to have GRE MRI before (or within 1 week) of starting best practice oral anticoagulant

Exclusion Criteria:

* Any MRI contraindications
* Previous use of oral anticoagulation
* Definite contra-indication to oral anticoagulation
* Serious head injury (resulting to loss of consciousness)

Study II: CROMIS-2 (ICH)

Inclusion criteria:

• Adult (>18y) patients treated at participating centres with confirmed ICH (confirmed on CT or MRI scans) with or without a history of anticoagulant use at the time of the ICH

Exclusion criteria:

* Known underlying structural cause for ICH (e.g arteriovenous malformation, tumour, cavernoma, intracranial aneurysm, haemorrhagic transformation of an infarct)
* Major head trauma (causing loss of consciousness and though to be sufficient to have caused the ICH) in previous 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study I: CROMIS-2 (AF) Prospective cohort study of patients anticoagulated after cardioembolic stroke Study I (AF): 1425 patients from UK centres. All eligible patients with first or recurrent ischaemic stroke and TIA in whom it is decided that best practice oral anticoagulant treatment is to be commenced.
  Study II (ICH): The investigators will recruit 600 patients treated at participating hospitals with ICH. Of these patients, 300 ICH cases will be related to anticoagulant use. The investigators will also recruit at least 300 ICH cases not related to anticoagulant use during the study period. Patients seen in outpatient clinics or from existing databases may also be recruited, at centres where these are available.
Sampling Method: Non-Probability Sample
Enrollment: 2490 (Actual)
Dates: Start 2011-08-04 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Symptomatic intracranial haemorrhage | 24 months
  Symptomatic intracranial haemorrhage (confirmed on brain imaging). Intracranial haemorrhage includes any bleeding within the skull, regardless of the site. The investigators will record the incidence of different haemorrhage subtypes (intracerebral, subdural, extradural, subarachnoid).
  This will be assessed using hospital records, General Practitioner (GP) follow up and National Health Service (NHS) information data system.

SECONDARY OUTCOMES:
Ischaemic stroke | 24 months
  Patient experiencing an ischaemic stroke during 2 year follow up.This will be assessed using hospital records, General Practitioner (GP) follow up and National Health Service (NHS) information data system.
Transient Ischaemic Attack (TIA) | 24 months
  Patient experiencing a TIA after recruitment during 2 year follow up.This will be assessed using hospital records, General Practitioner (GP) follow up and National Health Service (NHS) information data system.
Death | 24 months
  Patient death (of any cause). Assessed by General Practitioner (GP) follow up, recruiting hospital records and National Health Service (NHS) Information Centre data systems.
Any other major haemorrhagic events other than ICH | 24 months
  Prolonged epistaxis, cutaneous bruising, gastrointestinal bleeding, haematuria, muscle haematoma, haemarthrosis. Assessed by General Practitioner (GP) follow up, recruiting hospital records and National Health Service (NHS) Information Centre data systems.
Long term physical disability | 24 months
  Assessed by administering Modified Rankin Score (mRS) to patients at 6,12 and 24 months via patient questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: David Werring, Principal Investigator — UCL
Locations (1):
- UCL, London, United Kingdom

REFERENCES:
- [Derived] Seiffge DJ, Wilson D, Ambler G, Banerjee G, Hostettler IC, Houlden H, Shakeshaft C, Cohen H, Yousry TA, Al-Shahi Salman R, Lip G, Brown MM, Muir K, Jager HR, Werring DJ. Small vessel disease burden and intracerebral haemorrhage in patients taking oral anticoagulants. J Neurol Neurosurg Psychiatry. 2021 Mar 19;92(8):805-14. doi: 10.1136/jnnp-2020-325299. Online ahead of print. PMID 33741739
- [Derived] Hostettler IC, Schwarz G, Ambler G, Wilson D, Banerjee G, Seiffge DJ, Shakeshaft C, Lunawat S, Cohen H, Yousry TA, Al-Shahi Salman R, Lip GYH, Brown MM, Muir KW, Houlden H, Jager HR, Werring DJ; CROMIS-2 Collaborators. Cerebral Small Vessel Disease and Functional Outcome Prediction After Intracerebral Hemorrhage. Neurology. 2021 Apr 13;96(15):e1954-e1965. doi: 10.1212/WNL.0000000000011746. Epub 2021 Feb 24. PMID 33627495
- [Derived] Du H, Wilson D, Ambler G, Banerjee G, Shakeshaft C, Cohen H, Yousry T, Al-Shahi Salman R, Lip GYH, Houlden H, Brown MM, Muir KW, Jager HR, Werring DJ; Clinical Relevance of Microbleeds in Stroke (CROMIS-2) Collaborators. Small Vessel Disease and Ischemic Stroke Risk During Anticoagulation for Atrial Fibrillation After Cerebral Ischemia. Stroke. 2021 Jan;52(1):91-99. doi: 10.1161/STROKEAHA.120.029474. Epub 2020 Dec 7. PMID 33280548
- [Derived] Banerjee G, Wilson D, Ambler G, Hostettler IC, Shakeshaft C, Cohen H, Yousry T, Al-Shahi Salman R, Lip GYH, Houlden H, Muir KW, Brown MM, Jager HR, Werring DJ; CROMIS-2 collaborators. Longer term stroke risk in intracerebral haemorrhage survivors. J Neurol Neurosurg Psychiatry. 2020 Aug;91(8):840-845. doi: 10.1136/jnnp-2020-323079. Epub 2020 Jun 17. PMID 32554800
- [Derived] Banerjee G, Chan E, Ambler G, Wilson D, Cipolotti L, Shakeshaft C, Cohen H, Yousry T, Al-Shahi Salman R, Lip GYH, Muir KW, Brown MM, Jager HR, Werring DJ; CROMIS-2 Collaborators dagger; CROMIS-2 Collaborators<xref ref-type="author-note" rid="jah34726-note-1002"><sup>dagger</sup></xref>. Cognitive Impairment Before Atrial Fibrillation-Related Ischemic Events: Neuroimaging and Prognostic Associations. J Am Heart Assoc. 2020 Jan 7;9(1):e014537. doi: 10.1161/JAHA.119.014537. Epub 2020 Jan 4. PMID 31902325
- [Derived] Wilson D, Ambler G, Shakeshaft C, Banerjee G, Charidimou A, Seiffge D, White M, Cohen H, Yousry T, Salman R AS, Lip GYH, Muir K, Brown MM, Jager HR, Werring DJ; CROMIS-2 collaborators. Potential missed opportunities to prevent ischaemic stroke: prospective multicentre cohort study of atrial fibrillation-associated ischaemic stroke and TIA. BMJ Open. 2019 Jul 24;9(7):e028387. doi: 10.1136/bmjopen-2018-028387. PMID 31345970
- [Derived] Wilson D, Ambler G, Banerjee G, Shakeshaft C, Cohen H, Yousry TA, Al-Shahi Salman R, Lip GYH, Houlden H, Brown MM, Muir KW, Jager HR, Werring DJ; Clinical relevance of Microbleeds in Stroke (CROMIS-2) collaborators. Early versus late anticoagulation for ischaemic stroke associated with atrial fibrillation: multicentre cohort study. J Neurol Neurosurg Psychiatry. 2019 Mar;90(3):320-325. doi: 10.1136/jnnp-2018-318890. Epub 2018 Nov 19. PMID 30455404
- [Derived] Wilson D, Ambler G, Shakeshaft C, Brown MM, Charidimou A, Al-Shahi Salman R, Lip GYH, Cohen H, Banerjee G, Houlden H, White MJ, Yousry TA, Harkness K, Flossmann E, Smyth N, Shaw LJ, Warburton E, Muir KW, Jager HR, Werring DJ; CROMIS-2 collaborators. Cerebral microbleeds and intracranial haemorrhage risk in patients anticoagulated for atrial fibrillation after acute ischaemic stroke or transient ischaemic attack (CROMIS-2): a multicentre observational cohort study. Lancet Neurol. 2018 Jun;17(6):539-547. doi: 10.1016/S1474-4422(18)30145-5. Epub 2018 May 16. PMID 29778365
- [Derived] Banerjee G, Wilson D, Ambler G, Osei-Bonsu Appiah K, Shakeshaft C, Lunawat S, Cohen H, Yousry T Dr, Lip GYH, Muir KW, Brown MM, Al-Shahi Salman R, Jager HR, Werring DJ; CROMIS-2 Collaborators. Cognitive Impairment Before Intracerebral Hemorrhage Is Associated With Cerebral Amyloid Angiopathy. Stroke. 2018 Jan;49(1):40-45. doi: 10.1161/STROKEAHA.117.019409. Epub 2017 Dec 15. PMID 29247143
- [Derived] Charidimou A, Wilson D, Shakeshaft C, Ambler G, White M, Cohen H, Yousry T, Al-Shahi Salman R, Lip G, Houlden H, Jager HR, Brown MM, Werring DJ. The Clinical Relevance of Microbleeds in Stroke study (CROMIS-2): rationale, design, and methods. Int J Stroke. 2015 Oct;10 Suppl A100:155-61. doi: 10.1111/ijs.12569. Epub 2015 Aug 2. PMID 26235450